CLINICAL TRIAL: NCT04568161
Title: Chronic Effect of Doxorubicin and Cyclophosphamide on Neurovascular Control and Blood Pressure in Women in Adjuvant Treatment for Breast Neoplasia
Brief Title: Effect of Anthracyclines and Cyclophosphamide on Cardiovascular Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Universidade Federal Fluminense (Other); Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Breast Cancer Chemotherapy
Record Dates: First submitted 2020-08-26; First posted 2020-09-29 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Cardiotoxicity; Cardiovascular Disease; Neurovascular Disorder; Endothelial Disfunction; Breast Cancer
Keywords: Chemotherapy; Endothelial Disfunction; Muscle Sympathetic Nerve Activity; Blood Pressure
MeSH Terms: conditions — Cardiotoxicity; Cardiovascular Diseases; Breast Neoplasms | interventions — Heart Function Tests; Heart Rate; Blood Pressure; Anthracyclines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pre and post chemotherapy assessments (Experimental): The patients will be assessed before and after chemotherapy treatment.
  Interventions: Procedure: Physical Characteristics; Procedure: Muscular Sympathetic Nervous Activity; Diagnostic Test: Cardiac Function; Diagnostic Test: Heart rate; Diagnostic Test: Blood pressure; Diagnostic Test: Blood Assessments; Diagnostic Test: Muscle blood flow; Diagnostic Test: Endothelium-dependent vascular function; Diagnostic Test: Vascular intima-media thickness; Diagnostic Test: Physical Capacity; Drug: Anthracycline & Cyclophosphamide treatment scheme

INTERVENTIONS:
Procedure: Physical Characteristics — Body weight, height and waist circumference
Procedure: Muscular Sympathetic Nervous Activity — Microneurography technique.
Diagnostic Test: Cardiac Function — Echocardiography.
Diagnostic Test: Heart rate — Electrocardiography
Diagnostic Test: Blood pressure — Non-invasive photoplethysmography.
Diagnostic Test: Blood Assessments — Serum and Plasma will be extracted by centrifugation. Endothelial microparticles by flow cytometry Interleukin-6 and tumor necrosis factor α by ELISA, High-sensitive reactive serum C-reactive protein by immunoturbidimetric assay, NT- ProBNP According to Central Laboratory, Hospital das Clinicas, HCFMUSP, Faculdade de Medicina, Universidade de Sao Paulo. Endothelin-1 by immunoenzymatic method Nitric oxide by gas chemiluminescence Lipoperoxidation by fluorimetry Carbonyl by spectrophotometer, and Superoxide Dismutase (SOD) by colorimetry.
Diagnostic Test: Muscle blood flow — Venous occlusion plethysmography
Diagnostic Test: Endothelium-dependent vascular function — Brachial ultrasound
Diagnostic Test: Vascular intima-media thickness — Carotid ultrasound
Diagnostic Test: Physical Capacity — Cardiopulmonary exercise test
Drug: Anthracycline & Cyclophosphamide treatment scheme — Four session of intravenous (in bolus) infusion of doxorubicin 60mg/m2 and cyclophosphamide 600mg/m2 with an interval of 21 days between sessions.

SUMMARY:
The present study aims to investigate the chronic effect of treatment with doxorubicin and cyclophosphamide on neurovascular control and blood pressure in women undergoing adjuvant treatment for breast cancer.

DETAILED DESCRIPTION:
The development of new drugs and different adjuvant therapeutic regimens, based on the combination of anthracycline (A) and cyclophosphamide (C), have contributed greatly to improve survival rate in breast cancer patients. Despite the clinical benefits of this therapy, AC treatment can cause cardiovascular acute and chronic changes. In a recent investigation, we observed that an acute AC chemotherapy session increases sympathetic nervous activity and blood pressure in patients with breast cancer.

The present study aims to investigate the chronic effects of AC regimen on sympathetic nervous activity, peripheral vasoconstriction, endothelial microparticles and blood pressure, in women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stage II-III breast cancer
* starting adjuvant chemotherapy

Exclusion Criteria:

* metastatic disease,
* hypercholesterolemia, diabetes,
* hypertension,
* severe lymphedema,
* organic disorders (renal failure, heart failure and chronic liver disease),
* obesity (BMI> 30) and,
* who are under pharmacological treatment with statins, angiotensin-converting enzyme inhibitors, losartan potassium, beta blockers or antioxidants

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-09-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Muscle sympathetic nerve activity | 15-20 days after the end of AC regimen
  Change in muscular sympathetic nerve activity measured by microneurography

SECONDARY OUTCOMES:
Muscle blood flow | 15-20 days after the end of AC regimen
  Change in muscle blood flow measured by venous oclusion plethysmography
Blood Pressure | 15-20 days after the and of AC regimen
  Change in blood pressure measured by finometer
Physical capacity | 15-20 days after the end of AC regimen
  Change in physical capacity measured by cardiopulmonary exercise test
Cardiac Function Impairment | 15-20 days after the end of AC regimen
  Change in cardiac function measured by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E Negrao, PhD, Principal Investigator — Instituto do Coracao, HCFMUSP, Faculdade de Medicina, Universidade de Sao Paulo
Locations (1):
- Instituto do Coracao (InCor), Hospital das Clinicas HCFMUSP, Faculdade de Medicina, Universidade de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2019. CA Cancer J Clin. 2019 Jan;69(1):7-34. doi: 10.3322/caac.21551. Epub 2019 Jan 8. PMID 30620402
- [Background] Pai VB, Nahata MC. Cardiotoxicity of chemotherapeutic agents: incidence, treatment and prevention. Drug Saf. 2000 Apr;22(4):263-302. doi: 10.2165/00002018-200022040-00002. PMID 10789823
- [Background] Dolci A, Dominici R, Cardinale D, Sandri MT, Panteghini M. Biochemical markers for prediction of chemotherapy-induced cardiotoxicity: systematic review of the literature and recommendations for use. Am J Clin Pathol. 2008 Nov;130(5):688-95. doi: 10.1309/AJCPB66LRIIVMQDR. PMID 18854260
- [Background] Jensen BV, Skovsgaard T, Nielsen SL. Functional monitoring of anthracycline cardiotoxicity: a prospective, blinded, long-term observational study of outcome in 120 patients. Ann Oncol. 2002 May;13(5):699-709. doi: 10.1093/annonc/mdf132. PMID 12075737
- [Background] Sales ARK, Negrao MV, Testa L, Ferreira-Santos L, Groehs RVR, Carvalho B, Toschi-Dias E, Rocha NG, Laurindo FRM, Debbas V, Rondon MUPB, Mano MS, Hajjar LA, Hoff PMG, Filho RK, Negrao CE. Chemotherapy acutely impairs neurovascular and hemodynamic responses in women with breast cancer. Am J Physiol Heart Circ Physiol. 2019 Jul 1;317(7):H1-H12. doi: 10.1152/ajpheart.00756.2018. Epub 2019 Apr 19. PMID 31002284
- [Background] Soultati A, Mountzios G, Avgerinou C, Papaxoinis G, Pectasides D, Dimopoulos MA, Papadimitriou C. Endothelial vascular toxicity from chemotherapeutic agents: preclinical evidence and clinical implications. Cancer Treat Rev. 2012 Aug;38(5):473-83. doi: 10.1016/j.ctrv.2011.09.002. Epub 2011 Oct 6. PMID 21982720
- [Background] Laterza MC, de Matos LD, Trombetta IC, Braga AM, Roveda F, Alves MJ, Krieger EM, Negrao CE, Rondon MU. Exercise training restores baroreflex sensitivity in never-treated hypertensive patients. Hypertension. 2007 Jun;49(6):1298-306. doi: 10.1161/HYPERTENSIONAHA.106.085548. Epub 2007 Apr 16. PMID 17438307
- [Background] Barretto AC, Santos AC, Munhoz R, Rondon MU, Franco FG, Trombetta IC, Roveda F, de Matos LN, Braga AM, Middlekauff HR, Negrao CE. Increased muscle sympathetic nerve activity predicts mortality in heart failure patients. Int J Cardiol. 2009 Jul 10;135(3):302-7. doi: 10.1016/j.ijcard.2008.03.056. Epub 2008 Jun 26. PMID 18582965
- [Background] Jenkins NT, Padilla J, Boyle LJ, Credeur DP, Laughlin MH, Fadel PJ. Disturbed blood flow acutely induces activation and apoptosis of the human vascular endothelium. Hypertension. 2013 Mar;61(3):615-21. doi: 10.1161/HYPERTENSIONAHA.111.00561. Epub 2013 Jan 14. PMID 23319545
- [Background] Negrao CE, Rondon MU, Tinucci T, Alves MJ, Roveda F, Braga AM, Reis SF, Nastari L, Barretto AC, Krieger EM, Middlekauff HR. Abnormal neurovascular control during exercise is linked to heart failure severity. Am J Physiol Heart Circ Physiol. 2001 Mar;280(3):H1286-92. doi: 10.1152/ajpheart.2001.280.3.H1286. PMID 11179075
- [Background] Granger DL, Anstey NM, Miller WC, Weinberg JB. Measuring nitric oxide production in human clinical studies. Methods Enzymol. 1999;301:49-61. doi: 10.1016/s0076-6879(99)01068-x. No abstract available. PMID 9919553
- [Background] Kovachich GB, Mishra OP. Lipid peroxidation in rat brain cortical slices as measured by the thiobarbituric acid test. J Neurochem. 1980 Dec;35(6):1449-52. doi: 10.1111/j.1471-4159.1980.tb09022.x. PMID 7441260
- [Background] Thijssen DHJ, Bruno RM, van Mil ACCM, Holder SM, Faita F, Greyling A, Zock PL, Taddei S, Deanfield JE, Luscher T, Green DJ, Ghiadoni L. Expert consensus and evidence-based recommendations for the assessment of flow-mediated dilation in humans. Eur Heart J. 2019 Aug 7;40(30):2534-2547. doi: 10.1093/eurheartj/ehz350. PMID 31211361
- [Background] Abdel-Sayed S, Nussberger J, Aubert JF, Gohlke P, Brunner HR, Brakch N. Measurement of plasma endothelin-1 in experimental hypertension and in healthy subjects. Am J Hypertens. 2003 Jul;16(7):515-21. doi: 10.1016/s0895-7061(03)00903-8. PMID 12850383